CLINICAL TRIAL: NCT05132608
Title: Effect of a Social Media-based Health Education Program on Postnatal Care (PNC) Knowledge Among Pregnant Women Using Smartphones in Dhulikhel Hospital: a Randomized Controlled Trial
Brief Title: Effect of a Social Media-based Health Education Program on Postnatal Care (PNC) Knowledge Among Pregnant Women Using Smartphones in Dhulikhel Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kalpana Chaudhary, Principal Investigator, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 106/20
Record Dates: First submitted 2021-11-11; First posted 2021-11-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Unrecognized Condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media (Experimental): social media based health education program developed using Health belief model
  Interventions: Other: Social media-based Health education program
- Usual care (No Intervention): physical assessment of maternal and foetal wellbeing, screening, treatment, and receiving preventive measures

INTERVENTIONS:
Other: Social media-based Health education program — The social media-based health education program consist of 16 minute PNC video in Nepali language guided by Health Belief Model. The video provided general information on postnatal care including frequency, timing, and place providing postnatal care; danger signs of mother and newborn; different services provided at each PNC visit, and the importance of PNC visit. The researcher sent PNC videos through instant messaging (IM) software applications such as Viber, What's App, and Facebook messenger to the intervention group.
  Arms: Social Media

SUMMARY:
Its an interventional study conducted to assess the effect of social media-based health education program on PNC knowledge among pregnant women attending Dhulikhel hospital, Nepal.

DETAILED DESCRIPTION:
The study is a two-arm open-label randomized controlled trial conducted among literate pregnant visiting Dhulikhel hospital for ANC check-up. A computer-based program allocated 229 pregnant women owning smartphone with internet connectivity in a 1:1 ratio to either intervention (n=109) or usual care (n=120). The investigators assessed PNC knowledge in the participants by interviewing in-person or via phone; questionnaire was adopted from the previous study conducted to determine the knowledge of postnatal care among postpartum mothers in Asmara; that contained 20 knowledge questions with a maximum possible score of 61. The questionnaire was translated and pretested in Nepali, with the Cronbach alpa of 0.83. The intervention group received a 16 minutes video developed by using Health belief model via social media and the participants were reminded to view the video every week via telephone for a month. Control group received usual care. The primary outcome of the study was PNC knowledge score. The investigators utilized intent-to-treat analysis and measured the effect of the intervention on PNC knowledge score using linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* literate pregnant women
* owned a smartphone
* used social media (either What's App, Viber, or Facebook)
* had internet connectivity (WIFI or mobile data)

Exclusion Criteria:

• learning difficulties(dementia) or vision impairment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
PNC knowledge assessment | 3 months
  The investigators adopted knowledge assessment questionnaire from the hospital-based cross-sectional study conducted to determine the knowledge of postnatal care among postpartum mothers during discharge in maternity hospitals in Asmara

CONTACTS AND LOCATIONS:
Locations (1):
- Kalpana Chaudhary, Dhulikhel, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaye R, Schwaninger B, Hoffman D. Activator construction simplified. J Clin Orthod. 1979 Nov;13(11):773-8. No abstract available. PMID 298290
- [Derived] Chaudhary K, Nepal J, Shrestha K, Karmacharya M, Khadka D, Shrestha A, Shakya PR, Rawal S, Shrestha A. Effect of a social media-based health education program on postnatal care (PNC) knowledge among pregnant women using smartphones in Dhulikhel hospital: A randomized controlled trial. PLoS One. 2023 Jan 20;18(1):e0280622. doi: 10.1371/journal.pone.0280622. eCollection 2023. PMID 36662821